CLINICAL TRIAL: NCT04198805
Title: The Effect of Vitamin E and Docosahexaenoic Acid Ethyl Ester on Non-Alcoholic Fatty Liver Disease (NAFLD) - Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial (PUVENAFLD)
Brief Title: Vitamin E and DHA-EE on NAFLD - Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial (PUVENAFLD)
Acronym: PUVENAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naga P. Chalasani (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Naga P. Chalasani, Associate Dean of Research, Director of GI/Hepatology, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-1088
Record Dates: First submitted 2019-10-30; First posted 2019-12-13 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Fatty Liver; Non-Alcoholic Steatohepatitis
Keywords: Non-Alcoholic Fatty Liver Disease; Non-Alcoholic Fatty Liver; NAFL; NAFLD; Vitamin E; DHA
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Vitamin E; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vitamin E (1000 mg) (Active Comparator): Vitamin E (1000 mg) once daily for 6 months (1 capsule) and matching placebos (2 matched capsules) for 6 months.
  Interventions: Dietary Supplement: Vitamin E [(all-rac)-α-tocopheryl acetate]
- DHA EE (1.89 g) (Active Comparator): DHA EE (1.89 g) once daily for 6 months (2 capsules) and matching placebo for DHA EE (1 matched capsule for 6 months).
  Interventions: Dietary Supplement: Omega-3 fatty acid (DHA EE)
- DHA EE (1.89 g) and Vitamin E (1000 mg) (Active Comparator): DHA EE (1.89 g) once daily for 6 months and Vitamin E (1000 mg) once daily for 6 months.
  Interventions: Combination Product: Omega-3 fatty acid (DHA EE) & Vitamin E [(all-rac)-α-tocopheryl acetate]
- Placebo (Placebo Comparator): Matching soybean oil placebo (3 capsules) of all arms daily for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin E [(all-rac)-α-tocopheryl acetate] — Vitamin E (1000 mg) once daily for 6 months (1 capsule) and matching placebos (2 matched capsules) for 6 months
  Arms: Vitamin E (1000 mg)
Dietary Supplement: Omega-3 fatty acid (DHA EE) — DHA EE (1.89 g) once daily for 6 months (2 capsules) and matching placebo for DHA EE (1 matched capsule for 6 months)
  Arms: DHA EE (1.89 g)
Combination Product: Omega-3 fatty acid (DHA EE) & Vitamin E [(all-rac)-α-tocopheryl acetate] — DHA EE (1.89 g) once daily for 6 months and Vitamin E (1000 mg) once daily for 6 months
  Other Names: Vitamin E [(all-rac)-α-tocopheryl acetate]
  Arms: DHA EE (1.89 g) and Vitamin E (1000 mg)
Other: Placebo — Matching soybean placebo (3 capsules) of all arms daily for 6 months.
  Arms: Placebo

SUMMARY:
Multicenter, randomized, double-blinded, placebo-controlled clinical trial is focused on novel treatments for non-alcoholic fatty liver disease (NAFLD), the most common cause of chronic liver disease. The primary objective of the study is to determine the clinical efficacy and safety of Vitamin E [(all-rac)-α-tocopheryl acetate] and Omega-3 fatty acid (DHA EE) compared to placebo on reducing liver fat content in participants with NAFLD. There is currently no approved drug treatment for NAFLD or NASH. While several new targets are being evaluated, they are not sufficiently powered to provide definitive data. There is, therefore, a need for well-designed, appropriately powered efficacy (phase 2) trials to define the utility of newer therapies for NAFLD. The combination of Vitamin E and DHA may provide optimal benefit for patients with NAFLD due to their associated mechanisms of action, namely Vitamin E's antioxidant action, preventing lipid oxidation of long-chain fatty acids such as DHA and thus preventing the propagation of free radicals and ROS.

DETAILED DESCRIPTION:
Background information

Non-alcoholic fatty liver disease (NAFLD) is characterized by excessive fat accumulation in the liver and is defined by evidence of hepatic steatosis (via imaging or histology) and is not due to secondary liver fat accumulation from excessive alcohol consumption or hereditary disorders (e.g., Wilson's disease). NAFLD is most commonly associated with metabolic syndrome, consisting of obesity, insulin resistance, elevated blood pressure, and dyslipidemia. NAFLD is one of the most common causes of chronic liver disease, globally with a prevalence as high as 30% in Western countries. It includes a spectrum of diseases from steatosis to non-alcoholic steatohepatitis (NASH), liver fibrosis, cirrhosis, and hepatocellular carcinoma. Non-alcoholic fatty liver does not involve hepatocellular injury in the form of ballooning hepatocytes, whereas NASH is defined by steatosis, inflammation, and hepatocyte injury (ballooning) with or without fibrosis. The causes of NAFLD are likely due to a combination of genetic and physiologic factors, namely those that promote oxidative stress and inflammation such as metabolic syndrome, visceral adiposity, and changes in intestinal microbiota. NAFLD is significantly associated with increased risk of Type II Diabetes and cardiovascular disease and increased overall mortality compared to age-matched controls. There is currently no approved drug treatment for NAFLD or NASH. Dietary restrictions for weight loss and increased physical activity are the recommended therapies, albeit with limited success.

Investigational products

Vitamin E [(all-rac)-α-tocopheryl acetate]

Vitamin E is a fat-soluble vitamin that is synthesized naturally in plants in four tocopheryl forms: α, β, γ, and δ. All-rac-α-tocopheryl acetate has the highest biological activity in animal models, and it is the α-tocopheryl form that is used to prevent and treat Vitamin E deficiency in humans. Functionally, Vitamin E is an anti-oxidant and peroxyl radical scavenger. It is an inhibitor of lipid peroxidation and can also inhibit and modulate intracellular signaling molecules, e.g., protein kinase C, and nicotinamide adenine dinucleotide phosphate (NADPH) oxidase. α-tocopheryl regulates gene expression of several intracellular enzymes such as 5-lipoxygenase and cyclooxygenase and has anti-inflammatory activity (i.e., decreasing cytokine release and plasma C reactive protein). It is also known to inhibit platelet adhesion and aggregation. \

DHA Ethyl Ester

Long-chain polyunsaturated fatty acid (LC-PUFA), docosahexaenoic acid (DHA) is an essential omega-3 fatty acid for brain, eye and cardiovascular development and health. It significantly reduces triglycerides (TGs), lowers heart rate, lowers blood pressure, and reduces the risk of cardiac death by an overall 8%. Both DHA and eicosapentaenoic acid (EPA) have anti-thrombotic, anti-inflammatory, and anti-oxidative properties. As NAFLD patients are at significantly greater risk of cardiovascular disease and higher overall mortality, the cardioprotective effects of DHA are significant and may be beneficial in the NAFLD population.

Potential mechanisms for DHA's effects in NAFLD include the reduction of TG synthesis via activation of peroxisome proliferator-activated receptors (PPAR-α and γ), which accelerates fatty acid oxidation in liver mitochondria. DHA is also known to have an integral role in maintaining and improving cell membrane fluidity, as a fatty acid that is incorporated into the phospholipids of the membrane, thereby optimizing surface receptors and signal transduction pathways in liver cells. The anti-inflammatory role of DHA in NAFLD may be mediated through activation of adiponectin secretion through adults with NAFLD. MRI-PDFF is also an appropriate technique to diagnose and stage disease in those with metabolic syndrome and NAFLD. The clinical trial is designed to test the combination of Vitamin E and DHA against placebo, to demonstrate efficacy and safety.

Rationale for conducting the clinical study

The combination of Vitamin E and DHA has not been tested in previous clinical trials of adults with NAFLD. This combination may provide optimal benefit for patients with NAFLD due to their associated mechanisms of action, namely Vitamin E's antioxidant action, preventing lipid oxidation of long-chain fatty acids such as DHA and thus preventing the propagation of free radicals and ROS. Vitamin E's protection of LC-PUFA DHA, therefore, assists it in maintaining cell membrane stability and optimal signaling. Their combined anti-inflammatory effects (e.g., inhibiting pro-inflammatory cytokines, increasing adiponectin, and producing docosanoids to resolve inflammation) may also be efficacious for those with metabolic syndrome and NAFLD. The combination of Vitamin E and DHA will correctly be used in this study to determine if a reduction in liver fat occurs after six months of co-administration, using a magnetic resonance imaging (MRI) technique, proton density fat fraction (PDFF). PDFF imaging is non-invasive and highly sensitive to detect liver steatosis in patients with NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* ≥18 years of age
* A new diagnosis or reconfirmation of previously known fatty liver by imaging (ultrasound or CT or MRI), or by liver biopsy within ≤ 4 years
* Fibroscan CAP score >300db
* Hepatic fat fraction ≥12% by MRI PDFF
* ALT≥ 40 U/L
* eGFR/Creatinine Clearance ≥ 60ml/min
* Participants with previously diagnosed Type 2 diabetes (up to 50% of sample): they must either be taking anti-diabetic medications, or their fasting (>10 hours) glucose must be ≥ 100 mg/dL at the time of screening
* Stable weight (±5%) for at least 3 months
* Subjects willing and able to give written informed consent and to understand, to participant and to comply with the clinical study requirements.

Exclusion Criteria:

* Evidence of alternative causes of hepatic steatosis or other forms of chronic liver disease, e.g. Hep.B, Hep.C
* Evidence of acute Hepatitis A
* Serum ALT or AST ≥ 250 U/L
* Serum Alkaline Phosphatase > 2 ULN
* Total bilirubin > 2 ULN in the absence of Gilbert's Syndrome [In patients with Gilbert's Syndrome, direct bilirubin must not exceed 2 ULN]
* HbA1c≥9.5%
* Decompensated acute or chronic liver disease
* Clinical, imaging or histological evidence of cirrhosis
* Use of anti-NASH drugs (e.g. thiazolidinediones) in the 3 months prior to randomization
* Use of a non-stable dose of statins or fibrates in the 3 months prior to randomization
* Use of fish oil, algal oil or Krill oil supplements, drugs or foods fortified with omega-3s in the 2 months prior to randomization (>200mg DHA/d and/or >60mg EPA/d by FFQ)
* Known intolerance to vitamin E or DHA
* Malabsorption of Vit E (e.g. due to steatorrhea, chronic pancreatitis, severe cholestasis)
* Vitamin E supplementation of greater than 100 IU/day in the 3 months prior to randomization
* History of bariatric surgery (jejunoileal bypass or gastric weight loss surgery) or currently undergoing evaluation for bariatric surgery
* History of biliary diversion
* Known positivity for antibody to Human Immunodeficiency Virus (HIV)
* Patients with coagulopathy (PT ≥3 sec.from ULN), thrombocytopenia (<70K)
* Contraindication to MRI (implants, metal…)
* Active, serious medical disease or disease diagnosis of a life-expectancy less than 5 years
* Ongoing or recent alcohol consumption > 21 drinks (1 drink= 12 oz regular beer, or 5 oz wine, or 1.5 oz distilled spirits) per week in men and > 14 drinks per week in women as per subject self-report as part of medical history.
* Active substance abuse, such as oral, inhaled or injected illicit drugs (except marijuana), in the year prior to screening
* Women of childbearing potential: positive pregnancy test during screening or at randomization or unwillingness to use an effective form of birth control during the trial
* Women who are breastfeeding
* Any other condition which, in the opinion of the investigator would impede compliance or hinder completion of the study
* Subjects who are enrolled in an interventional clinical study or have received an investigational new drug or product within the last 30 days prior to screening
* Participants diagnosed with type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naga P. Chalasani, MD, Principal Investigator — Indiana University School of Medicine
Locations (15):
- United States (15):
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Integrity Clinical Research LLC, Doral, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Advanced Pharma CR LLC, Miami, Florida
  - Med-Care Research, Miami, Florida
  - Summit Clinical Research LLC, Athens, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - M3 Wake Research Associates, Raleigh, North Carolina
  - Centex Studies, Inc., Houston, Texas
  - Liver Specialists of Texas/Mt. Olympus Medical Research, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: April, 2024

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin E (1000 mg) | DHA EE (1.89 g) | DHA EE (1.89 g) and Vitamin E (1000 mg) | Placebo
Started | 34 | 34 | 67 | 70
Completed | 26 | 30 | 61 | 60
Not Completed | 8 | 4 | 6 | 10
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Early Termination | 8 | 4 | 6 | 9

BASELINE CHARACTERISTICS:
Population: Vitamin E ad DHA EE groups not consistent with participant workflow due to two subjects not completing MRI.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin E (1000 mg) | DHA EE (1.89 g) | DHA EE (1.89 g) and Vitamin E (1000 mg) | Placebo | Total
Number analyzed (Participants) | 33 | 34 | 66 | 70 | 203
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.3 (15.4) | 52.8 (12.8) | 50.0 (12.1) | 50.7 (12.6) | 50.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 35 | 34 | 108
  Male | 13 | 15 | 31 | 36 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 15 | 42 | 40 | 120
  Not Hispanic or Latino | 10 | 19 | 24 | 30 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 0 | 3 | 7 | 13
  White | 30 | 32 | 61 | 61 | 184
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 34 | 66 | 70 | 203

OUTCOME MEASURES:

1. Primary Outcome: Change in Hepatic Fat Fraction [%] Between of Vitamin E and DHA EE vs Placebo
Description: A change in liver fat content relative to baseline between Vitamin E and DHA EE vs placebo. This will be measured by MRI-PDFF at baseline and after 6 months of intervention (value at 6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: Participants analyzed varies from participant workflow due to inconsistencies in what was able to be collected at differing sites and timepoints
Measure: Mean (Standard Deviation); unit: Percentage of liver fat
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Placebo
Number analyzed (Participants) | 60 | 57
Percentage of liver fat | -6.8 (26.4) | -8.2 (18.2)

2. Secondary Outcome: Change in Hepatic Fat Fraction [%] Between Vitamin E vs Placebo Arm
Description: Change in liver fat content relative to baseline between Vitamin E vs placebo arm. This will be measured by MRI-PDFF at baseline and after 6 months of intervention (value at 6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of liver fat
Arm/Group | Vitamin E (1000 mg) | Placebo
Number analyzed (Participants) | 26 | 57
Percentage of liver fat | -10.4 (15.7) | -8.2 (18.2)

3. Secondary Outcome: Change in Hepatic Fat Fraction [%] Between DHA EE vs Placebo Arm
Description: Change in liver fat content relative to baseline between DHA EE vs placebo arm. This will be measured by MRI-PDFF at baseline and after 6 months of intervention (value at 6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of liver fat
Arm/Group | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 29 | 57
Percentage of liver fat | 2.2 (24.1) | -8.2 (18.2)

4. Secondary Outcome: Change After 6 Months of DHA EE and/ or Vitamin E Intervention in the Anthropometric Measure, Waist Circumference.
Description: Evaluation of baseline and 6 month measurements of waist circumference in the DHA EE and /or Vitamin E intervention over a 6 month period.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Groups:
- Vitamin E (1000 mg): Vitamin E (1000 mg) Vitamin E (1000 mg) once daily for 6 months (1 capsule) and matching placebos (2 matched capsules) for 6 months.
  Vitamin E [(all-rac)-α-tocopheryl acetate] Vitamin E (1000 mg) once daily for 6 months (1 capsule) and matching placebos (2 matched capsules) for 6 months
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 59 | 25 | 31 | 60
centimeters (cm) | 0.8 (6.5) | -0.5 (4.9) | -0.2 (6.0) | 0.8 (4.3)

5. Secondary Outcome: Change After 6 Months of DHA EE and /or Vitamin E Intervention in the Anthropometric Measure, Bodyweight.
Description: Evaluation of baseline and 6-month measurements of body weight in the DHA EE and /or Vitamin E intervention over a 6 month period.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 61 | 26 | 32 | 60
kilogram (kg) | 0.4 (3.7) | 0.5 (2.7) | 0.0 (4.1) | -0.0 (3.7)

6. Secondary Outcome: Change After 6 Months of DHA EE and/ or Vitamin E Intervention in the Anthropometric Measure, Waist-to-hip Ratio .
Description: Evaluation of baseline and 6-month measurements of waist-to-hip ratio (the circumference of the waist divided by the circumference of the hips) in the DHA EE and /or Vitamin E intervention over a 6 month period.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 59 | 25 | 31 | 59
ratio | 0.0 (0.0) | -0.0 (0.0) | 0.0 (0.0) | -0.0 (0.0)

7. Secondary Outcome: Change After 6 Months of DHA EE and/ or Vitamin E Intervention in the Anthropometric Measure, Body Mass Index (BMI)
Description: Evaluation of baseline and 6-month measurements of body mass index (BMI) in the DHA EE and /or Vitamin E intervention over a 6 month period.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 61 | 26 | 32 | 60
kg/m^2 | 0.1 (1.3) | 0.2 (1.0) | -0.0 (1.5) | -0.0 (1.3)

8. Secondary Outcome: Change in Insulin Levels to Determine Insulin Resistance
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ulU/mL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 58 | 24 | 31 | 61
ulU/mL | 4.7 (38.7) | -5.7 (47.8) | 9.9 (60.3) | 4.3 (43.9)

9. Secondary Outcome: Change in Liver Enzymes (ALT) in the DHA EE and /or Vitamin E Intervention Over a 6 Month Period.
Description: Evaluation of baseline and 6-month liver enzymes: alanine transaminase (ALT) in the DHA EE and /or Vitamin E intervention over a 6 month period value at (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 123 | 54 | 63 | 125
U/L | -4.6 (53.9) | -16.7 (30.5) | 7.0 (54.5) | -6.8 (32.3)

10. Secondary Outcome: Change in Liver Enzymes (AST) in the DHA EE and /or Vitamin E Intervention Over a 6 Month Period.
Description: Evaluation of baseline and 6-month liver enzymes: aspartate aminotransferase (AST) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 123 | 54 | 63 | 125
U/L | -1.4 (33.1) | -6.4 (25.1) | 2.9 (35.4) | -2.8 (22.5)

11. Secondary Outcome: Change in Liver Enzymes Bilirubin in the DHA EE and /or Vitamin E Intervention Over a 6 Month Period.
Description: Evaluation of baseline and 6-month liver enzymes: Bilirubin in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 123 | 54 | 63 | 125
mg/dL | 0.1 (0.2) | -0.0 (0.1) | -0.0 (0.2) | 0.1 (0.2)

12. Secondary Outcome: Liver Enzymes Alkaline Phosphatase in the DHA EE and /or Vitamin E Intervention Over a 6 Month Period.
Description: Evaluation of baseline and 6-month liver enzymes: Alkaline Phosphatase in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 123 | 54 | 63 | 126
U/L | -4.1 (15.6) | -0.4 (15.1) | 1.1 (11.2) | 2.5 (18.4)

13. Secondary Outcome: Change in Fibrosis-4 (FIB-4) Score
Description: The formula for FIB-4 is: Age ([yr] x AST [U/L]) / ((PLT [10(9)/L]) x (ALT [U/L])(1/2)). A value of FIB-4 below 1.30 is considered as low risk for advanced fibrosis; a value of FIB-4 over 2.67 is considered as high risk for advanced fibrosis
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 58 | 25 | 31 | 58
units on a scale | -0.1 (0.5) | -0.2 (0.5) | -0.1 (0.4) | -0.0 (0.5)

14. Secondary Outcome: Change in Plasma Vitamin E Concentration
Description: Evaluation of baseline and 6-month plasma Vitamin E concentration in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 61 | 25 | 31 | 62
ng/mL | 6972 (7217.1) | 9949 (10086.5) | 480.9 (2898.5) | 148.0 (2657.2)

15. Secondary Outcome: Change in Plasma DHA EE Concentration
Description: Evaluation of baseline and 6-month plasma DHA EE concentration in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 61 | 26 | 31 | 62
ug/mL | 41.6 (51.9) | 0.6 (24.9) | 52.8 (51.6) | -2.6 (17.5)

16. Secondary Outcome: Change in Lipid Profile (HDL-C)
Description: Evaluation of baseline and 6-month lipid profile (HDL-C) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 60 | 25 | 31 | 62
mg/dL | 1.7 (7.4) | 0.0 (9.5) | 2.4 (5.5) | 0.5 (10.2)

17. Secondary Outcome: Change in Lipid Profile (Low Density Lipoprotein (LDL-C))
Description: Evaluation of baseline and 6-month lipid profile (low density lipoprotein (LDL-C))in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 60 | 25 | 31 | 62
mg/dL | 9.9 (34.8) | 2.1 (27.3) | 19.4 (31.2) | 5.1 (25.7)

18. Secondary Outcome: Change in Lipid Profile (Triglycerides)
Description: Evaluation of baseline and 6-month lipid profile (TGs)in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 60 | 25 | 31 | 62
mg/dL | -23.1 (78.5) | 2.0 (107.3) | -6.6 (87.6) | -21.4 (93.9)

19. Secondary Outcome: Change in Lipid Profile (Oxidized LDL)
Description: Evaluation of baseline and 6-month lipid profile (oxidized LDL) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 60 | 25 | 31 | 62
U/L | 4.1 (13.4) | 5.3 (8.2) | 4.6 (13.2) | 0.5 (10.6)

20. Secondary Outcome: Change in Health Related Quality of Life Score (Short Form (SF-36))
Description: Evaluation of baseline and 6-month quality of life score (SF-36) in the DHA EE and /or Vitamin E intervention over a 6 month period (value at 6 months minus value at baseline). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 60 | 26 | 32 | 62
score on a scale
  Emotional Well-Being | -0.4 (12.6) | -1.9 (10.7) | 2.3 (13.0) | 0.5 (16.1)
  Energy/Fatigue | 0.5 (16.4) | 4.6 (11.1) | -1.4 (17.0) | 0.8 (17.5)
  General Health | -0.4 (15.2) | 0.4 (10.0) | 2.8 (14.7) | -2.7 (15.0)
  Pain | 0.4 (15.7) | 3.3 (9.7) | -0.8 (20.3) | 3.3 (18.7)
  Physical Functioning | -1.3 (21.5) | 1.5 (11.5) | 0.3 (18.0) | 0.8 (15.2)
  Role Limitations Due to Emotional Problems | -0.6 (33.9) | 7.7 (21.7) | 0.0 (22.4) | -3.2 (23.9)
  Role Limitations Due to Physical Health | -2.5 (27.1) | 5.8 (28.6) | 1.6 (35.9) | -4.4 (24.2)
  Social Functioning | 1.9 (16.4) | -1.0 (20.3) | 0.0 (16.8) | -1.6 (17.0)

21. Secondary Outcome: Change in Dietary Intake Levels of Long-chain Polyunsaturated Fatty Acids (LC-PUFA ) (i.e. DHA and EPA) as Measured by the Food Frequency Questionnaire (FFQ)
Description: Evaluation of baseline and 6-month dietary intake levels of LC-PUFA (i.e. DHA and EPA) as measured by the Food Frequency Questionnaire (FFQ)in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg per day
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 61 | 26 | 34 | 70
mg per day
  FFQ DHA | 2.3 (39.7) | 4.4 (14.9) | -0.7 (8.5) | -1.6 (12.5)
  FFQ EPA | 0.7 (19.7) | 2.4 (9.4) | -0.6 (4.8) | -0.8 (7.5)

22. Secondary Outcome: Change in Inflammatory Markers (Cytokeratin 18 (CK-18))
Description: Evaluation of baseline and 6-month inflammatory markers (cytokeratin 18) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 58 | 25 | 31 | 61
U/L | -17.7 (241.5) | -26.8 (215.7) | 37.3 (284.3) | 61 (15.1)

23. Secondary Outcome: Change in Inflammatory Markers (IL-1β)
Description: Evaluation of baseline and 6-month inflammatory markers (IL-1β) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 55 | 22 | 29 | 56
pg/mL | 0.0 (0.8) | -0.1 (1.1) | 0.2 (1.3) | -0.4 (2.9)

24. Secondary Outcome: Change in Inflammatory Markers (TNFα)
Description: Evaluation of baseline and 6-month inflammatory markers (TNFα) in the DHA EE and /or Vitamin E intervention over a 6 month period (6 months minus value at baseline).
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | DHA EE (1.89 g) and Vitamin E (1000 mg) | Vitamin E (1000 mg) | DHA EE (1.89 g) | Placebo
Number analyzed (Participants) | 55 | 22 | 29 | 56
pg/mL | -1.3 (3.4) | -0.2 (2.5) | -0.3 (2.9) | -0.5 (3.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitamin E (1000 mg) | DHA EE (1.89 g) | DHA EE (1.89 g) and Vitamin E (1000 mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/67 | 1/70
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 1/67 | 1/70
Other Adverse Events (participants affected / at risk) | 6/34 | 17/34 | 18/67 | 25/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (1000 mg) (N=34) | DHA EE (1.89 g) (N=34) | DHA EE (1.89 g) and Vitamin E (1000 mg) (N=67) | Placebo (N=70)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin E (1000 mg) (N=34) | DHA EE (1.89 g) (N=34) | DHA EE (1.89 g) and Vitamin E (1000 mg) (N=67) | Placebo (N=70)
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertonic Bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bell's Palsy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisioning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilic esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 3 (3)
abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diabetes mellitus type 2 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Migraine (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Liver function test increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Remnant hyperlipidemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasm skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Desmoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04198805/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT04198805/SAP_001.pdf